CLINICAL TRIAL: NCT06110481
Title: Bronchodilator Response To Inhaled Beta-2 Agonist and Anticholinergic Drugs in Children Born Preterm
Brief Title: Reversibility of Bronchial Obstruction in Children Born Preterm
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jana Tuková, Principal Investigator, Charles University, Czech Republic
Other Study IDs: CZ-VFN-PEDMET-BPD-001
Record Dates: First submitted 2023-09-11; First posted 2023-10-31 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-10

CONDITIONS: Bronchopulmonary Dysplasia; Chronic Lung Disease of Prematurity; Chronic Lung Disease of Newborn; Preterm Birth Complication; Bronchial Hyperreactivity; Bronchial Obstruction; Reversible Dilatation
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study aims to compare responses to different, commonly used inhaled bronchodilators in children born preterm with bronchial obstruction at spirometry. All children were diagnosed with Chronic Lung Disease of Immaturity (CLDI).

The main questions are:

* Is any inhaled bronchodilator or their combination generally superior in children with CLDI when assessing the reversibility of bronchial obstruction?
* Is there an individual difference in the effect of betamimetic, anticholinergic or their combination between children with CLDI?

Participants will:

* Come to our clinic in a stable state without acute infection and they will be randomly assigned to the first inhaled bronchodilator.
* They will then perform a spirometry test before and after the inhalation of the drug.
* This visit will repeat 3 times, each with a different bronchodilator (beta2agonist, anticholinergic and their combination).

DETAILED DESCRIPTION:
1. Outpatient follow-up - Parents are asked to sign the study consent form if the child meets the indication criteria. If the trial subject is not taking inhaled therapy, he/she may immediately continue to Check-up A. If the subject is taking short- or long-acting bronchodilators, these medications must be discontinued before each check-up and at the following intervals:

   * Short-acting β2 agonists (SABA) - 12 hours before the examination
   * Short-acting inhaled cholinergic antagonists (e.g. ipratropium bromide) - 12 hours before the examination
   * Long-acting inhaled betamimetics (long-acting β2 agonists, LABAs) - 48 hours before the examination
   * Long-acting muscarinic antagonists (LAMA) - one week before the examination
2. Check-up A - Baseline pre-interventional spirometry may be performed if the subject has no evidence of acute respiratory infection or has not had an acute respiratory infection two weeks previously. Otherwise, the examination should be rescheduled. Before baseline spirometry, the child is randomized to a dilatation test with inhaled salbutamol, ipratropium, or a combination of fenoterol/ipratropium. After a defined time interval (15 - 30 minutes), post-interventional spirometry follows.

   The subject is invited to attend Check-up B (which preferably follows 1 to 30 days after Check-up A, but no later than 3 months).
3. Check-up B - Baseline pre-interventional spirometry may be performed if the subject has no evidence of acute respiratory infection or has not had an acute respiratory infection two weeks previously. Otherwise, Check-up B should be rescheduled. Before baseline spirometry, another inhaled bronchodilator according to the preceding randomisation is applied. After a defined time interval (15 - 30 minutes), post-interventional spirometry follows. Resting spirometry with a dilatation test with another drug, the choice of which is guided by randomization, is performed.
4. Check-up C - Baseline pre-interventional spirometry may be performed if the subject has no evidence of acute respiratory infection or has not had an acute respiratory infection two weeks previously. Otherwise, Check-up C should be rescheduled. Baseline spirometry with the last bronchodilator not yet used is performed.

ELIGIBILITY:
Inclusion Criteria:

* children born preterm /before the 35th week of gestational age (35+0)/
* all subjects must have chronic lung disease of prematurity with bronchial obstruction, confirmed by spirometry
* subjects must be able to cooperate well in spirometry

Exclusion Criteria:

* The presence of another chronic respiratory disease (e.g., cystic fibrosis, primary ciliary dyskinesia, etc.). Asthma bronchiale is not an exclusion criterion, but subjects with CLDI combined with asthma bronchiale represent a specific subgroup of subjects and we perform a standardized therapeutic test with inhaled corticosteroids (ICS) administered for at least 12 weeks via a pressurized aerosol dispenser (pMDI) via an inhaler attachment before enrollement.
* Insufficient cooperation during spirometry.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children born preterm before 35+0 of gestational age (35+0) with chronic lung disease of prematurity with bronchial obstruction, confirmed by spirometry.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of spirometric parameters of bronchial obstruction in children born preterm to inhaled salbutamol, ipratropium bromide and combination of fenoterol with ipratropium bromide | baseline and post-interventional spirometry after 15-30 minutes (interval specific to bronchodilator) during three check-ups with min. time interval between check-ups 24 hours and max. 30 days
  Spirometric parameters of bronchial obstruction before and after inhaled application of bronchodilator during check-up. Three types of bronchodilators (salbutamol, ipratropium bromide and combined inhaler of fenoterol with ipratropium bromide) at three different check-ups will be tested with the order selected by randomisation.
  Z-score of baseline (pre-interventional) spirometric expiratory flow parameters (MMEF (l/s), MEF75 (l/s), MEF50 (l/s), MEF25 (l/s) retrieved from flow-volume curve compared to post-interventional z- scores of MMEF (l/s), MEF75 (l/s), MEF50 (l/s), MEF25 (l/s) values measured after a predefined time interval specific to bronchodilator (15-30 minutes). Four standardised doses of bronchodilators will be administered with metered-dose inhaler by spacer without a mask.
Change of spirometric parameters of lung volume in children born preterm to inhaled salbutamol, ipratropium bromide and combination of fenoterol with ipratropium bromide | baseline and post-interventional spirometry after 15-30 minutes (interval specific to bronchodilator) during three check-ups with min. time interval between check-ups 24 hours and max. 30 days
  Spirometric parameters of lung volume before and after inhaled application of bronchodilator during check-up. Three types of bronchodilators (salbutamol, ipratropium bromide and combined inhaler of fenoterol with ipratropium bromide) at three different check-ups will be tested with the order selected by randomisation.
  Z-score of baseline (pre-interventional) spirometric volume parameters FEV 0.5 (ml), FVC (ml) retrieved from flow-volume curve compared to post-interventional z- scores of FEV 0.5 (l), FVC (l) values measured after a predefined time interval specific to bronchodilator (15-30 minutes). Four standardised doses of bronchodilators will be administered with metered-dose inhaler by spacer without a mask.
Change of area under the flow-volume spirometric curve in children born preterm to inhaled salbutamol, ipratropium bromide and combination of fenoterol with ipratropium bromide | baseline and post-interventional spirometry after 15-30 minutes (interval specific to bronchodilator) during three check-ups with min. time interval between check-ups 24 hours and max. 30 days
  Complex spirometric parameter of area under the curve before and after inhaled application of bronchodilator during check-up. Three types of bronchodilators (salbutamol, ipratropium bromide and combined inhaler of fenoterol with ipratropium bromide) at three different check-ups will be tested with the order selected by randomisation.
  Z-score of baseline (pre-interventional) Aex (l*l/s) retrieved from flow-volume curve compared to post-interventional z- scores of Aex (l*l/s) values measured after a predefined time interval specific to bronchodilator (15-30 minutes). Four standardised doses of bronchodilators will be administered with metered-dose inhaler by spacer without a mask.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Tukova, MD,PhD, Principal Investigator — Charles University, Czech Republic First Faculty of Medicine, Prague
Locations (1):
- First faculty of Medicine, Charles university., Prague, Czechia